CLINICAL TRIAL: NCT03085706
Title: Transplantation of Autologous Peripheral Blood Mononuclear Cells in the Subarachnoid Space for Amyotrophic Lateral Sclerosis: a Safety Analysis of 14 Patients
Brief Title: Transplantation of Autologous Peripheral Blood Mononuclear Cells for Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Principal Investigator, Liu Jing, Chief Physician, The First Affiliated Hospital of Dalian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCKY2016-58
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: 14 patients conducted at the First Affiliated Hospital of Dalian Medical University, China were eligible if they had definite or probable sporadic amyotrophic lateral sclerosis (ALS).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PBMC autotransplantation (Experimental): Fourteen amyotrophic lateral sclerosis (ALS) patients are received peripheral blood mononuclear cell (PBMC) autotransplantation.
  Interventions: Biological: PBMC autotransplantation

INTERVENTIONS:
Biological: PBMC autotransplantation — Fourteen amyotrophic lateral sclerosis (ALS) patients are received peripheral blood mononuclear cell (PBMC) autotransplantation.

SUMMARY:
To assess the safety of peripheral blood mononuclear cell transplantation into the subarachnoid space for the treatment of amyotrophic lateral sclerosis.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a rapidly evolving, fatal neurodegenerative disease resulting from the degeneration of cortical, bulbar and spinal motor neurons. The disease progresses inexorably to death, usually because by failure of respiratory function, with a median duration of 3 years.

Recent clinical trials using various types of stem cells, including mesenchymal stromal cells, neural stem cells, and peripheral blood mononuclear cells (PBMCs), represent promising strategies for stem cell-based treatment in ALS. It has been demonstrated that the inflammation and neuronal death were reduced in ALS patients after bone marrow transplantation. In addition, the incidence of immune response was decreased by autologous transplantation of bone marrow cells in ALS patients. PBMCs are multi-potent stem cells that are very attractive for a cell therapy approach in ALS because of their plasticity and ability to provide the host tissue with growth factors or modulate the host immune system. PBMCs were used clinically and few adverse effects were attributed to their administration. Early clinical investigations indicated that the transplantation of autologous PBMCs into the dura is feasible in ALS patients; however, one study was limited to three patients and the other recruited eight patients. There are still many questions regarding the intrathecal transplantation of PBMCs for ALS. Therefore, a retrospective study was performed to assess further the safety and efficacy of the procedure and to test the impact of a cell therapy approach in ALS patients.

Statistical analysis Data, expressed as the mean ± SD, were analyzed using SPSS version 17.0 for Windows (SPSS Inc., Chicago, IL, USA). Statistical analyses were performed by paired sample t-test. A value of P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* all subjects had a verifiable diagnosis of ALS for 0.5 to 2 years based on a diagnosis using the Revised Criteria of the World Federation of Neurology. The grades of diagnosis were clinically definite ALS or clinically probable ALS;
* ALS was mild-to-moderate based on the ALS Functional Rating Scale-Revised. Electrophysiological features showed compound muscle action potential (CMAP) amplitude of motor nerve normal or mild declining;
* serum creatine kinase was normal or mild upper, less than 500 U/L.

Exclusion Criteria:

* use of any other investigational agent within 30 days before treatment;
* severe cardiac, pulmonary, hepatic or/and hematic disease;
* human immunodeficiency virus positivity or signs and symptoms consistent with human immunodeficiency virus infection;
* pregnant or nursing women;
* history of cancer with less than 5 years documentation of a disease-free state;
* history of anaphylactic reaction or hypersensitivity to granulocyte colony- stimulating factor (G-CSF);
* alcohol or drug abuse in recent 1 year;
* cannot understand or obey the rules of treatment;
* blood donor in recent 30 days.

Ages: 31 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
adverse events of autologous peripheral blood mononuclear cell mobilization | 1 week after operation
  To assess the safety of autologous peripheral blood mononuclear cell transplantation

SECONDARY OUTCOMES:
Functional independence measurement(FIM) | changes of preoperation and week 1, week 2, week 4, week 12 after operation
  To assess the self-care ability of daily living
Berg Balance Scale | changes of preoperation and week 1, week 2, week 4, week 12 after operation
  To assess the trunk balance capability and limb movement function
Dysarthria Assessment Scale | changes of preoperation and week 1, week 2, week 4, week 12 after operation
  To assess the progression of bulbar paralysis

CONTACTS AND LOCATIONS:
Overall Officials: Jing Liu, Ph.D., Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided